CLINICAL TRIAL: NCT02381483
Title: The Role of Vitamin A in Brown Fat Activity and Energy Metabolism
Brief Title: Vitamin A in Brown Fat Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Florian Kiefer, MD, PhD, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1032/2013
Record Dates: First submitted 2015-02-14; First posted 2015-03-06 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Brown Adipose Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lean (Experimental): Cold exposure
  Interventions: Other: Cold exposure
- Obese (Experimental): Cold exposure
  Interventions: Other: Cold exposure

INTERVENTIONS:
Other: Cold exposure

SUMMARY:
Vitamin A metabolites (retinoids) have shown to activate brown fat function in preclinical studies, however the role of retinoids in human brown fat physiology and energy metabolism remains elusive. This study aims to identify a possible association between retinoid metabolism, brown fat activity, and energy expenditure in lean and obese subjects by using FDG-PET-CT, PET-MR Scans and indirect calorimetry. Additionally we will analyze the genetic profile of white and brown neck fat biopsies at room temperature and cold conditions in a subset of the study participants. More detailed molecular studies (involving other potential browning markers) will also be performed in adipocytes derived from human SVC.

The optimal duration of cold exposure will be determined in a pilot study. Therefore subjects will be repeatedly exposed to cold and circulating retinoid levels and other plasma parameters will be measured at various time points.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 45 years.
* Body mass index (BMI) 18.5 - 24.9 kg/m2 (lean) or 30.0 - 38.0 kg/m2 (obese)

Exclusion Criteria:

* Endocrine (except hyperlipidemia), cardiovascular (except hypertension), liver, kidney, inflammatory bowel, rheumatic, oncologic disease or any other chronic condition.
* Medication for any of the above mentioned conditions.
* Pregnancy
* Metallic implants that are not MRI compatible

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-02; Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Correlation between retinol/retinol-binding protein concentrations and cold-induced brown fat acitivity | 6 years
  A possible association between serum retinol and retinol-binding protein concentrations and cold-induced brown fat activity in lean and obese subjects, respectively, will be analyzed.

SECONDARY OUTCOMES:
Analyses of potential BAT or browning markers in humans | 6 years
Association between BAT activity and energy expenditure | 6 years
Identification of new factors related to brown fat function | 6 years
  This is a very exploratory aim that involves a number of molecular tests. Therefore no single outcome measure can be defined here. Briefly, we will perform mRNA and miRNA analyses from BAT biopsies and plasma before and after cold exposure to identify new factors related to BAT function. Potential candidates will be tested in loss- or gain-of-function models in isolated human and/or murine adipocytes. In addition, the thermogenic effects of commercially available peptides, hormones, lipids, or steroid acids, will be tested in primary adipocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Kiefer, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Kulterer OC, Niederstaetter L, Herz CT, Haug AR, Bileck A, Pils D, Kautzky-Willer A, Gerner C, Kiefer FW. The Presence of Active Brown Adipose Tissue Determines Cold-Induced Energy Expenditure and Oxylipin Profiles in Humans. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa183. doi: 10.1210/clinem/dgaa183. PMID 32343312